CLINICAL TRIAL: NCT00303355
Title: An Evaluation of the Utility of Clinical Examination for the Measurement of Jugular Venous Pulse in Critically Ill Patients.
Brief Title: Measurement of Jugular Venous Pulse in Critically Ill Patients.
Status: Terminated | Type: Observational
Why Stopped: Study completed
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 11803B
Record Dates: First submitted 2006-03-14; First posted 2006-03-16 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Jugular Venous Pulse Measurement in Critically Ill Patients
Keywords: jugular venous pulse

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
To assess the utility of clinical bedside examination for the measurement of jugular venous pulse in critically ill patients.

DETAILED DESCRIPTION:
Procedures: All patients with central venous catheters (CVP) will undergo physical examination of the jugular veins, while blinded to the actual CVP measured from the catheter. Clinicians with various experience levels (attending physician, fellow, resident physician, 4th year medical student) will participate.

The following clinical data will be obtained: Demographic data such as age, sex, weight and diagnosis will be collected. Each clinician's bedside CVP will be recorded from the bedside monitor. Clinicians will be blinded to bedside monitor.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the ICU who have existing central venous catheters.

Exclusion Criteria:

* Patients admitted to the ICU who do not have existing central venous catheters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2002-09; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: J P Kress, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Vinayak AG, Levitt J, Gehlbach B, Pohlman AS, Hall JB, Kress JP. Usefulness of the external jugular vein examination in detecting abnormal central venous pressure in critically ill patients. Arch Intern Med. 2006 Oct 23;166(19):2132-7. doi: 10.1001/archinte.166.19.2132. PMID 17060544